CLINICAL TRIAL: NCT00344227
Title: Prospective Optical Coherence Tomography (OCT) Imaging of Patients With Neovascular Age-Related Macular Degeneration (AMD) Treated With Intra-Ocular Lucentis™ (Ranibizumab): PrONTO Study
Brief Title: Prospective OCT Study With Lucentis for Neovascular AMD (PrONTO Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-FVF3102s; FVF3102s
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2006-06-26 (Estimated); Status verified 2006-06

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: neovascularization; age-related macular degeneration; vascular endothelial growth factor (VEGF); antigen-binding fragment (Fab); antiangiogenesis; optical coherence tomography (OCT)
MeSH Terms: conditions — Neovascularization, Pathologic; Macular Degeneration; Fanconi Anemia, Complementation Group B | interventions — Ranibizumab

INTERVENTIONS:
Drug: Lucentis (Ranibizumab)

SUMMARY:
The PrONTO Study was designed to evaluate the response of neovascular age-related macular degeneration (AMD) patients to intravitreal Lucentis using Optical Coherence Tomography (OCT) imaging. OCT was then used to determine the need for retreatment after 3 monthly injections of Lucentis. Patients would be followed for 2 years.

DETAILED DESCRIPTION:
This is a Phase II, open-label study of intravitreally administered ranibizumab (LucentisTM). Ranibizumab is an anti Vascular Endothelial Growth Factor (VEGF) antibody fragment. Approximately 40 subjects with primary or recurrent subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD) will be enrolled. Lesion types included will be minimally classic or occult (predominatly occult) lesions or predominantly classic CNV, if the patient had received prior PDT (no more than 3 treatments). The study will be conducted at one study site.

After reading the informed consent and having all their questions answered by the investigator and the coordinator, the subjects will sign the informed consent prior to participation in a screening period that could last up to 28 days to determine eligibility. Fluorescein angiograms (FA) will be used to determine CNV classification for study eligibility. In addition, optical coherence tomography (OCT) will provide information on retinal thickness, subretinal fluid and sub retinal pigment epithelium fluid for study eligibility. Fluorescein angiograms and OCT will be evaluated by the Bascom Palmer Reading Center. OCT images will be evaluated primarily using the standard Zeiss Stratus OCT software (Vers. 3) to determine study eligibility and retinal thickness. Proprietary software algorithms in development and not yet validated by the FDA may be used for future data analysis but will not be included in the intial data analysis. The angiographic features that will permit participation will include evidence of CNV with subfoveal involvement of the lesion. The OCT features that will permit participation will include retinal thickness (macular edema) ≥300 microns, subretinal fluid ≥100 microns in thickness, or a detachment of the retinal pigment epithelium ≥100 microns in thickness. ETDRS visual acuity measurements must be between 20/40 and 20/400.

All eligible subjects will receive a ranibizumab dose of 500 micrograms at baseline and every 30 days thereafter for the first two months. ETDRS visual acuity testing and OCT measurements will be performed prior to injection. After each of the first 3 injections (baseline, Month-1, and Month-2), patients will return on post-injection days 1, 2, 4, 7, and 14. OCT measurements will be performed at those visits. ETDRS visual acuity measurements will be performed on each injection day and on post-injection day #14. At the Month-3 follow-up exam and thereafter, if the vision is stable or improved (stable visual acuity score= ±4 letters; improved visual acuity score ≥ 5 letters) from the previous visit, and there is no evidence of leakage from CNV as determined by fluorescein angiography and OCT, then no injection will performed. If the previous criteria are not met, then injections are continued monthly until these criteria are fulfilled. At that point, no further injections will be given until there is evidence of recurrent CNV.

Enrolled subjects, who did not have predominantly classic CNV at baseline but converted to predominantly classic CNV within the study, will be offered veteporfin photodynamic therapy (PDT). If a patient receives PDT, there will be no injection of ranibizumab at that visit, and the next injection of ranibizumab will not be performed for at least 1 month. Patients will continue in the study and receive additional PDT at 3 months intervals if needed. There will alaways be at least a 1 month separation between PDT and the subsequent ranibizumab injection.

The following criteria will need to be fulfilled to resume injections. There will need to be evidence of vision loss ≥ 5 letters associated with evidence of leakage from CNV as determined by OCT or fluorescein angiography, or a new-onset macular hemorrhage, or new onset classic CNV, or an increase in central macular thickness ≥ 100 microns.

Only one eye will be chosen as the "study eye". Only the study eye will receive intravitreal injections of ranibizumab.

Subjects will have scheduled monthly visits throughout the study for the evaluation of safety and efficacy. Subjects will have the first treatment of a ranibizumab injection by the injecting physician on Day 0 and will undergo retinal analysis by OCT on Days 1, 2, 4, 7 and 14 after the first 3 study treatments. At subsequent visits (every month [30±7 days]), the subject will have a safety evaluation by the evaluating physician prior to possible retreatment. After months 3 subjects will be contacted by the site personnel 2 days (±1 day) after each study treatment to elicit reports of any decrease in vision, eye pain, unusual redness, or any other new ocular symptoms; subjects will also be asked whether they have taken the prescribed self-administered post-injection antimicrobials. During the first 3 months, these questions will be asked when they return to clinic. Every 3 months, subjects will undergo fluorescein angiography and color fundus photography. Subjects will have a final safety visit at Month 24.

Fundus photography and fluorescein angiography will be performed at baseline and at months 3, 6, 12, 18, and 24. Additional fluorescein angiography will be performed at visits when it is decided that injections should be stopped (if continued past Month-3) or be resumed due to decreased vision and possible evidence of leakage from CNV. Optical coherence tomography will be performed at baseline and on days 1, 2, 4, 7, 14 after each of the first 3 injections. Since preliminary data suggest that OCT imaging can detect the earliest manifestations of recurrent CNV, all patients will be monitored once injections have been stopped using monthly ophthalmologic exams, ETDRS visual acuity measurements, and OCT imaging at each monthly follow-up visit up to month 24.

ELIGIBILITY:
Inclusion Criteria:

* • All subjects must meet the following criteria to be eligible for study entry: Signed informed consent

  * Age greater than 50 years
  * Active primary or recurrent subfoveal lesions with CNV secondary to AMD in the study eye, as defined in Table 1
  * Lesions with occult CNV or with some classic CNV component are permissible. However, if predominantly classic CNV (well-demarcated hyperfluorescence boundaries in the early phase of the fluorescein angiogram) is present, the patient must have had prior PDT (up to 3 previous photodynamic therapy treatments).
  * The OCT features that will permit participation will include retinal thickness (macular edema) ≥300 microns, subretinal fluid ≥100 microns in thickness, or a detachment of the retinal pigment epithelium ≥100 microns in thickness
  * The total area of CNV (including both classic and occult components) encompassed within the lesion must be ≥ 50% of the total lesion area
  * The total lesion area must be <12 disc areas (DA) in size.
  * Best corrected visual acuity, using ETDRS charts, of 20/40 to 20/400 (Snellen equivalent) in the study eye
  * Only one eye will be assessed in the study. If both eyes are eligible, the one with the better acuity will be selected for treatment and study unless, based on medical reasons, the investigator deems the other eye the more appropriate candidate for treatment and study.

Exclusion Criteria:

* • Prior treatment with verteporfin, external-beam radiation therapy, or transpupillary thermotherapy in the study eye (predominantly classic CNV can however only be included if the subject had up to 3 prior PDT treatments)

  * Treatment with verteporfin in the non-study eye less than 7 days preceding Day 0
  * Previous participation in a clinical trial (for either eye) involving anti angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)
  * Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye
  * Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding Day 0
  * History of vitrectomy, submacular surgery, or other surgical intervention for AMD in the study eye
  * Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals) Lesion Characteristics
  * Subfoveal fibrosis or atrophy in the study eye
  * CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-08; Study Completion 2007-04

PRIMARY OUTCOMES:
Mean Visual Acuity
Total number of treatments

SECONDARY OUTCOMES:
Time to decrease of OCT central retinal thickness
Time to improved visual acuity
Proportion gaining 3 lines of vision
Proportion stable or improved
Frequency of Retreatment

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Rosenfeld, MD, PhD, Principal Investigator — Bascom Palmer Eye Institute
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

REFERENCES:
- [Derived] Lalwani GA, Rosenfeld PJ, Fung AE, Dubovy SR, Michels S, Feuer W, Davis JL, Flynn HW Jr, Esquiabro M. A variable-dosing regimen with intravitreal ranibizumab for neovascular age-related macular degeneration: year 2 of the PrONTO Study. Am J Ophthalmol. 2009 Jul;148(1):43-58.e1. doi: 10.1016/j.ajo.2009.01.024. Epub 2009 Apr 18. PMID 19376495